CLINICAL TRIAL: NCT00786994
Title: Randomized, Multicenter, Double Blind Study to Compare the Efficacy and Tolerability of Oleogel-S-10 for 3 Month Versus Placebo Only in Patients With Mild to Moderate Actinic Keratoses Located at the Face and Head Oleogel-S-10 in Actinic Keratoses Trial
Brief Title: The Efficacy and Tolerability of Oleogel-S-10 in Patients With Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Birken AG (Industry)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAK-08
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Oleogel-S10 100 mg/g ointment for three months once a day (54 patients)
  Interventions: Drug: Oleogel-S10 100 mg/g
- 2 (Experimental): Oleogel-S10 100 mg/g ointment for three months twice a day (54 patients)
  Interventions: Drug: Oleogel-S10 100 mg/g
- 3 (Placebo Comparator): Placebo (petroleum jelly) for three months once a day (27 patients)
  Interventions: Drug: Placebo (petroleum jelly)
- 4 (Placebo Comparator): Placebo (petroleum jelly) for three months twice a day (27 patients)
  Interventions: Drug: Placebo (petroleum jelly)

INTERVENTIONS:
Drug: Oleogel-S10 100 mg/g — topical use once or twice daily
  Arms: 1; 2
Drug: Placebo (petroleum jelly) — topical use once or twice daily
  Other Names: Vaseline
  Arms: 3; 4

SUMMARY:
In this study the impact of Oleogel-S-10 versus placebo on actinic keratoses over a treatment period of 3 months will be tested. Additionally, once and twice daily applications are tested.

DETAILED DESCRIPTION:
Oleogel-S-10 has shown efficacy and was well tolerated in two previous clinical trials. In the second open label phase II trial the efficacy of Oleogel-S-10 alone was similar compared to a more invasive treatment with cryotherapy. Response rates of 85% with a clear-ance of more than 75 % of the lesions of the patients treated with Oleogel-S-10 over three months were reported. These encouraging results led to the present randomized, multicenter, double blind phase II trial. The efficacy of the treatment shall be tested in a double blind placebo controlled (petroleum jelly) fashion in order to obtain more reliable results for the planning of a phase III study.

ELIGIBILITY:
Inclusion Criteria:

* At least two mild to moderate actinic keratoses located at the facial skin or the head (except lips)
* Actinic keratoses with a diameter of 0,5 - 2 cm,

  * that are definitely distinguished from other lesions and display a minimum distance of 0,5 cm to neighbored lesions
  * that are evaluated as histopathological grade 1 to 3
* histologically proven AK within three months before study entry
* prepared and able to give written informed consent
* ≥ 18 years of age
* In case of females: postmenopause defined as

  * natural menopause with menses > 1 year ago
  * serum FSH (> 20 IU/l) and E2 levels in the postmenopausal range or
  * patients who had bilateral oophorectomy
* prepared and comply with all study requirements, including the following:

  * application of Oleogel-S10 on the treatment area once or twice a day
  * 4 clinic visits during the pre-study, treatment, post-treatment, and follow-up period
  * pre- and post-treatment biopsy for histological confirmation (of clearance) of AK-diagnosis
* Representative histologic slide and tissue block were shipped

Exclusion Criteria:

* Active immunosuppressive therapy
* data of clinically significant, unstable, cardiovascular or hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities or diseases Note: Patients with clinically stable medical conditions including, but not limited to, controlled hypertension, diabetes mellitus type II, hypercholesterolemia, or osteoarthritis will be allowed to enter the study
* known allergies to any excipient in the study drug
* any dermatological disease and/or condition in the treatment or surrounding area (3 cm distances from treatment area) that may be exacerbated by treatment with Oleogel-S-10 or cause difficulty with examination
* active chemical dependency or alcoholism, as assessed by the investigator
* pregnant and lactating women
* currently participating in another clinical study or have completed another clinical study with an investigational drug within the past 30 days
* received topical treatment at the treatment area with diclofenac gel, imiquimod or 5-FU within a time period of 1 month
* Concomitant existence of non-treated (non-excised) basal cell carcinoma, squamous cell carcinoma or malignant melanoma
* Invasive tumors within the treatment area, e.g.: merkel cell carcinoma, squamous cell carcinoma, basal cell carcinoma, the latter is accepted if completely surgically removed Note: A biopsy of any lesion within the treatment or surrounding area suggestive of malignancy should be performed at the pre-study screening visit. If invasive SCC or other malignant conditions are confirmed within the treatment area, the patient will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof. Dr., Principal Investigator — Universitätshautklinik Tübingen
Locations (6):
- Germany (4):
  - Charité University Hospital, Berlin
  - University Dermatology Hospital, Freiburg im Breisgau
  - University Dermatology Hospital, Tübingen
  - Dermatology practice, Wuppertal
- Greece (2):
  - National University, "Andreas Syggros" Skin & Venereal Diseases Hospital, Athens
  - University Dermatology Hospital, Heraklion

REFERENCES:
- [Result] Pflugfelder A, Andonov E, Weide B, Dirschka T, Schempp C, Stockfleth E, Stratigos A, Kruger-Krasagakis S, Bauer J, Garbe C, Eigentler TK. Lack of activity of betulin-based Oleogel-S10 in the treatment of actinic keratoses: a randomized, multicentre, placebo-controlled double-blind phase II trial. Br J Dermatol. 2015 Apr;172(4):926-32. doi: 10.1111/bjd.13342. Epub 2015 Feb 25. PMID 25124939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 165 patients were recruited.
Pre-assignment Details: 157 patients were evaluated in the ITT population. 8 of 165 recruited patients were excluded from ITT evaluation due to a deviation from the inclusion and exclusion criteria. For safety evaluations, all 165 patients had received treatment with study medication and all 165 patients were assessed for adverse events.
Groups:
- A - Oleogel-S10 Once Daily: Oleogel-S10 ointment for three months once a day (54 patients)
  Oleogel-S10: topical use once or twice daily
- B - Oleogel-S10 Twice Daily: Oleogel-S10 vehicle for three months twice a day (54 patients)
  Oleogel-S10: topical use once or twice daily
- C - Placebo Once Daily: Placebo (petroleum jelly) for three months once a day (27 patients)
  Placebo (petroleum jelly)
- D - Placebo Twice Daily: Placebo (petroleum jelly) for three months twice a day (27 patients)
  Placebo (petroleum jelly)
Period: Overall Study
Arm/Group | A - Oleogel-S10 Once Daily | B - Oleogel-S10 Twice Daily | C - Placebo Once Daily | D - Placebo Twice Daily
Started | 57 | 54 | 26 | 28
ITT | 53 | 51 | 25 | 28
Completed | 47 | 39 | 24 | 22
Not Completed | 10 | 15 | 2 | 6

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Oleogel-S10 Once Daily | B - Oleogel-S10 Twice Daily | C - Placebo Once Daily | D - Placebo Twice Daily | Total
Number analyzed (Participants) | 53 | 51 | 25 | 28 | 157
Age, Continuous [Median (Full Range); unit: years] | 72 [61 to 88] | 74 [56 to 85] | 69 [57 to 81] | 72 [51 to 83] | 72 [51 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 20 | 25 | 128
  Male | 12 | 9 | 5 | 3 | 29
Actinic keratosis baseline severity index [Number; unit: participants]
  Mild | 22 | 18 | 9 | 13 | 62
  Moderate | 31 | 33 | 16 | 15 | 95
Histopathological grading [Number; unit: participants]
  Grade I | 9 | 4 | 2 | 2 | 17
  Grade II | 11 | 10 | 4 | 12 | 37
  Grade III | 32 | 36 | 19 | 13 | 100
  not done | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response of the Marker Actinic Keratosis, Defined as Histologically Complete or Partial Clearance.
Description: Objective response of the marker actinic keratosis, defined as histologically complete or partial clearance (partial clearance = down-grading in Cockerell-classification). The marker actinic keratosis is defined as an initially selected lesion within the target area that will be used for final biopsy.
  The Cockerell classification refers to a single lesion, graded as the presence of atypical cells in the lower third of the epidermis (grade I), involvement of at least the lower two-thirds (grade II) or atypical keratinocytic proliferation in the entire epidermis (grade III). Thus a down-grading from a higher Cockerell grade (e.g., III) to a lower Cockerell grade (e.g., I) represents a positive outcome and treatment success.
Time Frame: 18 weeks
Measure: Number; unit: participants
Groups:
- A - Oleogel-S10 Once Daily: Oleogel-S10 ointment for three months once a day
  Oleogel-S10: topical use once or twice daily
- B - Oleogel-S10 Twice Daily: Oleogel-S10 vehicle for three months twice a day
  Oleogel-S10: topical use once or twice daily
- C/D - Placebo Once or Twice Daily: Placebo (petroleum jelly) for three months once or twice a day
  Placebo (petroleum jelly)
Arm/Group | A - Oleogel-S10 Once Daily | B - Oleogel-S10 Twice Daily | C/D - Placebo Once or Twice Daily
Number analyzed (Participants) | 47 | 39 | 46
participants
  Success: Downgrading or clearance | 22 | 17 | 19
  Failure: No downgrading or clearance | 25 | 22 | 27
Statistical Analysis 1: Comparison: A - Oleogel-S10 Once Daily vs C/D - Placebo Once or Twice Daily; A vs C/D; Test type: Superiority or Other; p = 0.60, Mantel Haenszel
Statistical Analysis 2: Comparison: B - Oleogel-S10 Twice Daily vs C/D - Placebo Once or Twice Daily; B vs. C/D; Test type: Superiority or Other; p = 0.83, Mantel Haenszel

ADVERSE EVENTS:
Time Frame: Treatment period of 18 weeks: Visits at 0, 6, 12 and 18 weeks
Groups:
- C - Placebo Once Daily: Placebo (petroleum jelly) for three months once a day
  Placebo (petroleum jelly)
- D - Placebo Twice Daily: Placebo (petroleum jelly) for three months twice a day
  Placebo (petroleum jelly)
Arm/Group | A - Oleogel-S10 Once Daily | B - Oleogel-S10 Twice Daily | C - Placebo Once Daily | D - Placebo Twice Daily
Serious Adverse Events (participants affected / at risk) | 2/57 | 3/54 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 3/57 | 7/54 | 3/26 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Oleogel-S10 Once Daily (N=57) | B - Oleogel-S10 Twice Daily (N=54) | C - Placebo Once Daily (N=26) | D - Placebo Twice Daily (N=28)
Fracture of rib (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolaps of intervertebral disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Oleogel-S10 Once Daily (N=57) | B - Oleogel-S10 Twice Daily (N=54) | C - Placebo Once Daily (N=26) | D - Placebo Twice Daily (N=28)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Flu-like syndrome (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough / upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement on publication prior to disclosure